CLINICAL TRIAL: NCT06577376
Title: A Multicenter, Open-label Phase I/II Clinical Study to Evaluate the Safety and Efficacy of Simmitinib or Irinotecan Liposomes Combined With DP303c Injection in the Treatment of HER2 Expressing Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma
Brief Title: A PhaseⅠ/Ⅱ Study of Simmitinib or Irinotecan Liposomes Combined With DP303c in Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Runshi Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSA1501-010
Record Dates: First submitted 2024-08-21; First posted 2024-08-29 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Localized Advanced or Metastatic Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma; Expressing Human Epidermal Growth Factor Receptor-2 (HER-2); Disease Progression After Receiving at Least One and at Most Two Lines of Systemic Treatment in the Past
MeSH Terms: interventions — Paclitaxel; Docetaxel; Irinotecan

STUDY DESIGN:
Intervention Model Description: In the dose escalation phase, a "3+3" approach is used to explore the safety and tolerability of subjects, and in the randomized controlled phase, the efficacy of different combination doses is explored
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- DP303c injection, dose level 1, Q3W + simmitinib tablets, dose level 1, D1-D21, Q4W (Experimental): DP303c injection, dose level 1, intravenous drip, Q3W + simmitinib tablets, dose level 1, oral, QD, taken for 3 weeks, discontinued for 1 week, Q4W
  Interventions: Drug: DP303c; Drug: Simmitinib tablets
- DP303c injection, dose level 1, Q3W + simmitinib tablets, dose level 2, D1-D21, Q4W (Experimental): DP303c injection, dose level 1, intravenous drip, Q3W + simmitinib tablets, dose level 2, oral, QD, taken for 3 weeks, discontinued for 1 week, Q4W
  Interventions: Drug: DP303c; Drug: Simmitinib tablets
- DP303c injection, dose level 1, Q2W + simmitinib tablets, dose level 2, D1-D21, Q4W (Experimental): DP303c injection, dose level 1, intravenous drip, Q2W + simmitinib tablets, dose level 2, oral, QD, taken for 3 weeks, discontinued for 1 week, Q4W
  Interventions: Drug: DP303c; Drug: Simmitinib tablets
- DP303c injection, dose level 2, Q3W + simmitinib tablets, dose level 2, D1-D21, Q4W (Experimental): DP303c injection, dose level 2, intravenous drip, Q3W + simmitinib tablets, dose level 2, oral, QD, taken for 3 weeks, discontinued for 1 week, Q4W
  Interventions: Drug: DP303c; Drug: Simmitinib tablets
- DP303c RP2D + irinotecan liposomes RP2D (Experimental)
  Interventions: Drug: DP303c; Drug: Irinotecan liposomes
- Single agent chemotherapy chosen by researchers (Active Comparator): Single agent chemotherapy chosen by researchers: paclitaxel, docetaxel, or irinotecan
  Interventions: Drug: Paclitaxel or docetaxel or irinotecan

INTERVENTIONS:
Drug: DP303c — DP303c is an antibody conjugate drug (ADC), composed of one anti-HER2 monoclonal antibody coupled to one MMAE via an enzyme specific linker
  Arms: DP303c RP2D + irinotecan liposomes RP2D; DP303c injection, dose level 1, Q2W + simmitinib tablets, dose level 2, D1-D21, Q4W; DP303c injection, dose level 1, Q3W + simmitinib tablets, dose level 1, D1-D21, Q4W; DP303c injection, dose level 1, Q3W + simmitinib tablets, dose level 2, D1-D21, Q4W; DP303c injection, dose level 2, Q3W + simmitinib tablets, dose level 2, D1-D21, Q4W
Drug: Simmitinib tablets — A novel small molecule inhibitor targeting fibroblast growth factor receptor (FGFR), vascular endothelial growth factor receptor (VEGFR2, KDR), and colony-stimulating factor 1 receptor (CSF-1R)
  Arms: DP303c injection, dose level 1, Q2W + simmitinib tablets, dose level 2, D1-D21, Q4W; DP303c injection, dose level 1, Q3W + simmitinib tablets, dose level 1, D1-D21, Q4W; DP303c injection, dose level 1, Q3W + simmitinib tablets, dose level 2, D1-D21, Q4W; DP303c injection, dose level 2, Q3W + simmitinib tablets, dose level 2, D1-D21, Q4W
Drug: Irinotecan liposomes — A chemotherapy
  Arms: DP303c RP2D + irinotecan liposomes RP2D
Drug: Paclitaxel or docetaxel or irinotecan — Paclitaxel or docetaxel or irinotecan is used as a control.
  Arms: Single agent chemotherapy chosen by researchers

SUMMARY:
This study is divided into two parts: Cohort 1 and Cohort 2. Cohort 1 includes the dose escalation phase of DP303c combined with simmitinib, as well as the randomized controlled trial (RCT) phase of DP303c combined with simmitinib; Cohort 2 includes dose escalation/dose extension of DP303c combined with irinotecan liposomes, as well as RCT stage of DP303c combined with irinotecan liposomes.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18-75 (including) years old; 2. Gastric adenocarcinoma or gastroesophageal junction adenocarcinoma diagnosed by histology or cytology; 3. Disease progression after receiving one or two lines of systemic treatment in the past (first-line treatment must be platinum/fluorouracil combination chemotherapy with or without immune checkpoint inhibitors); 4. There should be at least one measurable lesion according to the response evaluation criteria in solid tumors (RECIST v1.1),; 5. HER2 expression status: 2+ to 3+(applicable to Cohort 1) or 1+(applicable to Cohort 2); 6. Adequate organ or bone marrow function

Exclusion Criteria:

* *Eligibility Criteria:

Inclusion Criteria:

1. Aged 18-75 (including) years old;
2. Gastric adenocarcinoma or gastroesophageal junction adenocarcinoma diagnosed by histology or cytology;
3. Disease progression after receiving one or two lines of systemic treatment in the past (first-line treatment must be platinum/fluorouracil combination chemotherapy with or without immune checkpoint inhibitors);
4. There should be at least one measurable lesion according to the response evaluation criteria in solid tumors (RECIST v1.1),;
5. HER2 expression status: 2+ to 3+(applicable to Cohort 1) or 1+(applicable to Cohort 2);
6. Adequate organ or bone marrow function

Exclusion Criteria:

1. Patients who have experienced toxicity during previous treatment with trastuzumab or trastuzumab biosimilars, resulting in permanent discontinuation of trastuzumab or trastuzumab biosimilars;
2. Patients with a history of allergies to any component of DP303c and deemed severe by the researchers
3. There is uncontrolled serosal fluid accumulation that requires frequent drainage or medical intervention;
4. Active leptomeningeal disease or uncontrolled CNS metastasis;
5. Has a history of serious cardiovascular and cerebrovascular diseases;
6. There was a peripheral neuropathy of grade ≥ 2 (refer to NCI CTCAE 5.0) prior to enrollment;
7. History of gastrointestinal perforation and/or fistula within 6 months of first use of medication;
8. Inability to swallow medication orally or presence of clinically significant gastrointestinal diseases;
9. Urine protein ≥++ and 24-hour urine protein quantification>1.0 g during screening period;
10. There are eye diseases that require intervention, such as corneal diseases, retinal diseases, or active eye infections;
11. Used CYP3A4 strong inhibitors or CYP3A4 strong inducers 14 days before the first medication ;
12. Used UGT1A1 strong inhibitor before first medication and wash-off period is less than 5 half-lives.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-08-26 (Estimated); Primary Completion 2026-08-26 (Estimated); Study Completion 2027-08-26 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) occurrence and incidence | Up to approximately 36 months after the first participant is enrolled
Adverse events (AE) occurrence and incidence | Up to approximately 36 months after the first participant is enrolled
Objective response rate (ORR) per RECIST 1.1 | Up to approximately 36 months after the first participant is enrolled
Serious adverse events (SAE) occurrence and incidence | Up to approximately 36 months after the first participant is enrolled

SECONDARY OUTCOMES:
Disease control rate (DCR) per RECIST 1.1 | Up to approximately 36 months after the first participant is enrolled
Duration of response (DoR) per RECIST 1.1 | Up to approximately 36 months after the first participant is enrolled
Progression free survival (PFS) per RECIST 1.1 | Up to approximately 36 months after the first participant is enrolled
Overall survival(OS) | Up to approximately 36 months after the first participant is enrolled
Blood drug concentration of DP303c | Up to approximately 36 months after the first participant is enrolled
Blood concentration of total anti-DP303c antibody | Up to approximately 36 months after the first participant is enrolled
Positive incidence of anti-DP303c antibody (ADA) | Up to approximately 36 months after the first participant is enrolled
HER2 expression level | Up to approximately 36 months after the first participant is enrolled
Blood concentration of simmitinib | Up to approximately 36 months after the first participant is enrolled